CLINICAL TRIAL: NCT00658762
Title: A Phase 3, Randomized, Double-Blind, Parallel Group, 10-Week Placebo Controlled Fixed Dose Study of PD 0332334 and Paroxetine Evaluating the Efficacy and Safety of PD 0332334 for the Treatment of Generalized Anxiety Disorder
Brief Title: A 10-week Study Evaluating the Efficacy and Safety of PD 0332334 for the Treatment of Generalized Anxiety Disorder (3)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A5361020
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PD 0332334 225 mg BID (Experimental)
  Interventions: Drug: PD 0332334
- PD 0332334 300 mg BID (Experimental)
  Interventions: Drug: PD 0332334
- Paroxetine 20 mg q am (Active Comparator)
  Interventions: Drug: paroxetine
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PD 0332334 — Capsules, oral, 225 mg BID, 8 weeks, with 2 week taper
  Other Names: imagabalin
  Arms: PD 0332334 225 mg BID
Drug: PD 0332334 — Capsules, oral, 300 mg BID, 8 weeks, with 2 week taper
  Arms: PD 0332334 300 mg BID
Drug: paroxetine — Capsules, oral, 20 mg q am, 8 weeks, with 2 week taper
  Arms: Paroxetine 20 mg q am
Drug: Placebo — Capsules, oral, BID, 8 weeks, with 2 week taper
  Arms: Placebo BID

SUMMARY:
This is a 10-week trial that evaluates the efficacy and safety of PD 0332334 in subjects ages 18 and older with generalized anxiety disorder.

DETAILED DESCRIPTION:
Termination reason: On February 23rd 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GAD (Diagnostic and Statistical Manual-IV [DSM-IV], 300.02) as established by the clinician (psychiatrist or licensed clinical psychologist) who has interviewed the subject using all sources of data including the Mini International Neuropsychiatric Interview (MINI) for DSM-IV Axis I disorders and other clinical information. Subjects with specific phobia(s) (as defined in DSM-IV) or dysthymic disorder will be allowed in the study.
* Subjects must have a HAM-A total score >/= 20 at the screening (V1) and randomization (V2) visits. Subjects must also have a Covi Anxiety Scale score of >/= 9 and a Raskin Depression Scale score </= 7 at the Screening (V1) visit to ensure predominance of anxiety symptoms over depression symptoms.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, pancreatic, neurologic, active infections, immunological, or allergic disease (including drug allergies).
* Any of the following current (within the past 6 months through the present) DSM-IV Axis I diagnoses: Major depressive disorder; Obsessive compulsive disorder; Panic disorder; Agoraphobia; Posttraumatic stress disorder; Anorexia; Bulimia; Caffeine-induced anxiety disorder; Alcohol or substance abuse or dependence unless in full remission for at least 6 months; Social anxiety disorder.
* Any of the following past or current DSM-IV Axis I diagnoses: Schizophrenia; Psychotic disorder; Delirium, dementia, amnestic and other clinically significant cognitive disorders; Bipolar or schizoaffective disorder; Cyclothymic disorder; Dissociative disorders.
* Antisocial or borderline personality disorder.
* Serious suicidal risk per the clinical investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in HAM-A total score at Week 8 | 8 weeks
To assess the safety and tolerability of PD 0332334 in subjects with GAD | 8 weeks with taper

SECONDARY OUTCOMES:
Response rate on the HAM-A at Week 1 and Week 8 | 8 weeks
Remission rate based on the HAM-A at Week 8 | 8 weeks
Change from Baseline in the somatic subscale score of the HAM-A (item 7-13) at Week 8 | 8 weeks
Change from Baseline to Week 8 on the Medical Outcomes Study - Sleep Scale subscales | 8 weeks
Worsening and improvement (from Baseline to Week 8) on the Changes in Sexual Functioning Questionnaire (CSFQ). | 8 weeks
Change from Baseline to Week 8 on the Sheehan Disability Scale (SDS) total score | 8 weeks
Change from Baseline in the HAM-A total score at Weeks 1, 2, 4 and 6) | 6 weeks
Response rate on the PGI-C at Week 8 | 8 weeks
Response rate on the CGI-I at Week 1 and Week 8 | 8 weeks
Change from Baseline to Week 8 on the Medical Outcomes Study Sleep Scale (MOS-SS) Sleep Disturbance Score | 8 weeks
Average (across the Week 1, 2, 4, 6 and 8 visits) HAM-A Change from Baseline score | 8 weeks
Change from Baseline to Days 2-8 and Weeks 2, 4, 6 and 8 on the GA-VAS (diary) | 8 weeks
The "Week 1 Sustained Responser" rate based on the HAM-A | 8 weeks
Change from Baseline in the psychic subscale score of the HAM-A (Items 1-6 and 14) at Week 8. | 8 weeks
Change from Baseline to Days 2-8 and Weeks 2, 4, 6, 8 on the DAS-A (total score) | 8 weeks
Change from Baseline to Week 8 in the Q-Les-Q General Activities Score | 8 weeks
Change from Baseline to Week 1 on the Medical Outcomes Study Sleep Scale (MOS-SS) Sleep Disturbance Score | 1 week
Change from Baseline in the 17-item HAM-D total score at Weeks 1, 2, 4, and 8 | 8 weeks
Change from Baseline in CGI-S at Week 8 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (25):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Wildomar, California
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Greenwood, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Salem, Oregon
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Woodstock, Vermont
- Pfizer Investigational Site, Budapest, Hungary

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361020&StudyName=A%2010-week%20Study%20Evaluating%20the%20Efficacy%20and%20Safety%20of%20PD%200332334%20for%20the%20Treatment%20of%20Generalized%20Anxiety%20Disorder%20%283%29